CLINICAL TRIAL: NCT00114413
Title: Asthma Control Evaluation (ACE): A Biomarker-Based Approach to Improving Asthma Control and Mechanistic Studies (DAIT ICAC-02)
Brief Title: Evaluation of an Asthma Treatment Strategy Based on Exhaled Nitric Oxide Measurements in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ICAC-01/DAIT ICAC-02
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: Exhaled Nitric Oxide; Lung; Urban Health; Child; Adolescent
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference Strategy (Active Comparator): Participants in the reference strategy group will undergo the eNO procedure but will follow NAEPP guidelines alone for asthma treatment without eNO measurements for the rest of the study.
  Interventions: Drug: Inhaled corticosteroids
- Biomarker Strategy (Experimental): Participants in the biomarker strategy group will follow NAEPP treatment guidelines, as well as eNO measurements, to determine asthma treatment at each study visit.
  Interventions: Drug: Inhaled corticosteroids; Procedure: eNO measurement

INTERVENTIONS:
Drug: Inhaled corticosteroids — Used for both regular asthma control and as a rescue inhaler
Procedure: eNO measurement — measured by Aerocrine® NIOX device
  Arms: Biomarker Strategy

SUMMARY:
The purpose of ICAC-01 is to determine whether an asthma treatment strategy that measures exhaled nitric oxide (eNO) to indicate disease progression is more effective in treating asthma symptoms when combined with existing asthma treatment guidelines than treatment using the guidelines alone.

DETAILED DESCRIPTION:
Over the past two decades, the prevalence of asthma has dramatically increased in many parts of the world. The current National Asthma Education and Prevention Program (NAEPP) identifies inhaled corticosteroids (ICS) as the preferred long-term control therapy for all forms of persistent asthma. However, there is still a significant proportion of patients with persistent asthma who are not receiving ICS therapy or do not follow their treatment plan. Individualized asthma treatment plans are needed. The use of biomarkers, in addition to NAEPP guidelines, may help enhance the level of asthma assessment, guide medication regimens, and improve overall asthma control. This study will determine whether NAEPP-recommended treatment, combined with eNO measurement, is more effective in reducing asthma symptoms than NAEPP-recommended treatment alone. ICAC-01 will last 46 weeks and will comprise 8 study visits.

ICAC-01 also includes a mechanistic sub-study (ICAC-02). Its primary objective is to determine whether "highly sensitized", compared to "weakly sensitized" asthmatic subjects have more severe asthma, as defined by the levels at randomization to the completion of ICAC-01. To address the primary objective of ICAC-02, the study will include all the participants enrolled in ICAC-01 with dust mite-, cockroach- and/or alternaria-specific IgE levels within certain parameters.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma made by a doctor over a year prior to study entry OR symptoms have been present more than a year if the diagnosis was made less than a year prior to study entry
* Have symptoms consistent with persistent asthma OR have evidence of uncontrolled disease. More information on this criterion can be found in the DAIT ICAC-01 protocol.
* Currently reside in a pre-selected area containing at least 20% of households below the U.S. government poverty level
* Do not smoke and have not used smokeless tobacco products in the year prior to study entry
* Able to perform eNO measurement procedures and spirometry at study screening
* Parent or guardian willing to provide informed consent, if applicable
* History of clinical varicella (chicken pox) or have received varicella vaccine
* Planning to stay in the area for the next 12 months
* Primary language is English. Spanish speakers may enroll at centers with Spanish-speaking staff.
* Parent or guardian primarily speaks English (or Spanish at centers with Spanish-speaking staff), for participants with parent or guardian providing informed consent
* Willing to allow the study physician to manage disease for the duration of the study
* Willing to change asthma medications in order to follow the protocol

Exclusion Criteria:

* Adherence to controller medication between Visits 1 and 2 is less than 25%. More information on this criterion can be found in the DAIT ICAC-01 protocol.
* Determined to have mild intermittent asthma at Visit 1
* Have had a life-threatening asthma exacerbation requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure in the 5 years prior to study entry
* Have significant medical illnesses other than asthma. More information on this criterion can be found in the DAIT ICAC-01 protocol.
* Unable to use a metered-dose inhaler for administration of a beta-agonist rescue medication or a dry powder inhaler for the administration of asthma controller regimens
* Known hypersensitivity to any medications commonly used for the treatment of asthma
* Have not completed a home evaluation within 4 weeks of study screening
* Currently participating in another asthma-related drug or intervention study, or have participated in another asthma-related drug or intervention study in the month prior to study entry
* Does not sleep at least 4 nights per week in one home
* Lives with a foster parent (not applicable if patient is able to provide informed consent)
* Does not have access to a phone
* Requires certain medications. More information on this criterion can be found in the DAIT ICAC-01 protocol.
* Urine cotinine level above 100 ng/ml at study screening
* Pregnant or breastfeeding

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 547 (Actual)
Dates: Start 2004-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Mean maximum symptom days per 2 weeks, as assessed by questionnaire | At Visits 3 and 8

SECONDARY OUTCOMES:
Days with wheeze | Throughout study
Days of slowed down or discontinued physical activities due to asthma | Throughout study
Nights awoken due to asthma | Throughout study
Days on which plans were changed due to asthma | Throughout study
Days missed school/work due to asthma | Throughout study
Unscheduled office/clinic visit due to asthma | Throughout study
Emergency room/urgent care center due to asthma | Throughout study
Hospitalization due to asthma | Throughout study
Number of asthma exacerbations requiring prednisone or prednisone equivalent | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: William Busse, MD, Principal Investigator — University of Wisconsin, Madison
Locations (12):
- United States (12):
  - University of Arizona (DAIT-ICAC-01/02), Tucson, Arizona
  - National Jewish Medical and Research Center (DAIT-ICAC-01/02), Denver, Colorado
  - Howard University, Washington D.C., District of Columbia
  - Children's Memorial Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai (DAIT-ICAC-01/02), New York, New York
  - Rho Federal System Division, Inc- data coordinating center, Chapel Hill, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Texas Southwestern (DAIT-ICAC-01/02), Dallas, Texas
  - University of Wisconsin-an administrative site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Reid DW, Johns DP, Feltis B, Ward C, Walters EH. Exhaled nitric oxide continues to reflect airway hyperresponsiveness and disease activity in inhaled corticosteroid-treated adult asthmatic patients. Respirology. 2003 Dec;8(4):479-86. doi: 10.1046/j.1440-1843.2003.00495.x. PMID 14629652
- [Background] Strunk RC, Szefler SJ, Phillips BR, Zeiger RS, Chinchilli VM, Larsen G, Hodgdon K, Morgan W, Sorkness CA, Lemanske RF Jr; Childhood Asthma Research and Education Network of the National Heart, Lung, and Blood Institute. Relationship of exhaled nitric oxide to clinical and inflammatory markers of persistent asthma in children. J Allergy Clin Immunol. 2003 Nov;112(5):883-92. doi: 10.1016/j.jaci.2003.08.014. PMID 14610474
- [Background] Langley SJ, Goldthorpe S, Custovic A, Woodcock A. Relationship among pulmonary function, bronchial reactivity, and exhaled nitric oxide in a large group of asthmatic patients. Ann Allergy Asthma Immunol. 2003 Oct;91(4):398-404. doi: 10.1016/S1081-1206(10)61688-2. PMID 14582820
- [Background] Jones SL, Herbison P, Cowan JO, Flannery EM, Hancox RJ, McLachlan CR, Taylor DR. Exhaled NO and assessment of anti-inflammatory effects of inhaled steroid: dose-response relationship. Eur Respir J. 2002 Sep;20(3):601-8. doi: 10.1183/09031936.02.00285302. PMID 12358335
- [Result] Szefler SJ, Mitchell H, Sorkness CA, Gergen PJ, O'Connor GT, Morgan WJ, Kattan M, Pongracic JA, Teach SJ, Bloomberg GR, Eggleston PA, Gruchalla RS, Kercsmar CM, Liu AH, Wildfire JJ, Curry MD, Busse WW. Management of asthma based on exhaled nitric oxide in addition to guideline-based treatment for inner-city adolescents and young adults: a randomised controlled trial. Lancet. 2008 Sep 20;372(9643):1065-72. doi: 10.1016/S0140-6736(08)61448-8. PMID 18805335
- [Result] Arroyave WD, Rabito FA, Carlson JC, Sever ML, Lefante J. Asthma severity, not asthma control, is worse in atopic compared with nonatopic adolescents with asthma. Ann Allergy Asthma Immunol. 2016 Jan;116(1):18-25. doi: 10.1016/j.anai.2015.10.015. Epub 2015 Nov 7. PMID 26560898
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY210 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY210 — ImmPort study identifier is SDY210. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts and is available to the Public.
- Available data/document: Study Protocol: SDY210 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY210 — ImmPort study identifier is SDY210. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts and is available to the Public.
- Available data/document: Study summary and schematic, -design, adverse event(s), -interventions,-medications, -demographics, and -files.: SDY210 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY210 — ImmPort study identifier is SDY210. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts and is available to the Public.